CLINICAL TRIAL: NCT02011178
Title: Prevention of Microvascular Complications in Overweight Diabetics With Surgery or Best Medicine; a Prospectivee, Randomized, Multicenter Study
Brief Title: Prevention of Microvascular Complications in Overweight Diabetics With Surgery or Best Medicine
Acronym: PROMISE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects have been enrolled
Sponsor: Karolinska Institutet (Other)
Collaborators: St. Claraspital AG (Other)
Responsible Party: Principal Investigator, Anders Thorell, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1530-31
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal medical treatment and surgery (Active Comparator): In the study 50 obese patients with CKD 3 andT2DM will be treated using the European Association for Study of Diabetes protocol in combination with RYGB surgery.
  Interventions: Procedure: Optimal medical treatment and surgery
- Optimal medical treatment (Other): In the study 50 obese patients with CKD 3 andT2DM will be treated using the European Association for Study of Diabetes protocol
  Interventions: Procedure: Optimal medical treatment

INTERVENTIONS:
Procedure: Optimal medical treatment and surgery
  Arms: Optimal medical treatment and surgery
Procedure: Optimal medical treatment
  Arms: Optimal medical treatment

SUMMARY:
Background: Diabetic kidney disease (DKD) is chronic and often progresses to kidney failure,heart disease and premature death. Unfortunately, the best medical therapies available for DKD today are ultimately unable to prevent its progression, especially in obese patients.Surgical rerouting of food within the gut with a gastric bypass operation (RYGB), improves diabetes and some of its complications.

The investigators propose to investigate whether RYGB in combination with best medical therapy in patients with DKD and obesity prevent further deterioration of kidney function over a 3 years follow up period.

Study design: This is an international collaboration with leading centres in Sweden and Switzerland in which100 obese type 2 diabetic patients with established DKD will volunteer to be randomly assigned to receive best medical therapy with RYGB or best medical therapy without surgery. Participants will be 18-65 years with type 2 diabetes and impaired kidney function. Yearly measurements of kidney function will then be done over a period of 3 years as a primary outcome to determine whether differences in DKD can be detectable. The study will also examine and compare a) safety of the interventions, b) the health economic impact on direct healthcare costs and Quality of Life in patients as well as c) the value of a new marker of DKD in determining which patients are most likely to benefit from surgery.

Overall the study will strengthen the evidence base guiding clinical decisions about the usefulness of RYGB as an add on therapy to best medical therapy in stopping progressive DKD in patients with obesity and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* • BMI 28 - 35 kg/m2

  * Age: 18-65 years, with T2DM
  * Estimated glomerular filtration rate (eGFR; by MDRD) between 30 and 60mL/min/1.73m2
  * Urine albumin creatinine ratio (ACR) of at least 30mg/g (microalbuminuria) in first void urine on two separate days.

Exclusion Criteria:

* • Type 1 diabetes or a positive GAD antibody test

  * Known renal artery stenosis
  * Renal impairment for reasons unrelated to diabetes
  * Suspicion of glomerulonephritis as determined by urine sediment (>10 erythrocytes/visual field)
  * Post-renal obstruction diagnosed by ultrasound
  * Severe retinopathy (defined as high-risk proliferative diabetic retinopathy and severe visual loss according to the "Early Treatment Diabetic Retinopathy Study Severity Scale")
  * Severe DKD (CKD 4 or 5, requirement of renal replacement therapy such as dialysis or kidney transplantation)
  * Severe neuropathy (peripheral neuropathy stage 3)
  * Unacceptably high risk for general anesthesia
  * Prior extensive intra-abdominal surgery making laparoscopy complicated
  * Myocardial infarction, cerebrovascular accident, transient ischemic attack, coronary-artery bypass grafting or percutaneous transluminal coronary angioplasty within the previous 6 months
  * Cardiac failure (NYHA stage > 2)
  * Inability to stop smoking prior to inclusion
  * Pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate | Three years after intervention
  Renal function measurement by Iohexol clearance

SECONDARY OUTCOMES:
Microvascular kidney damage | 3 years after intervention
  Microvascular kidney damage measured by Albumin/Creatinine Ratio
Glycaemic control | 3 years after intervention
  HbA1c and fasting plasma glucose measurements . Five day continuous glucose monitoring
peripheral nervous system function | 3 years after intervention
  Michigan Neuropathy Screening Instrument (MNSI) score, which includes two separate assessments: a lower extremity examination that includes inspection of the feet to identify deformities, dry skin, calluses, infection, fissure, or ulcers, and assessment of vibratory sensation and ankle reflexes
autonomic nervous system function | 3 years after intervention
  Autonomic neuropathy will be assessed with the RR intervals on ECG during deep breathing test
diabetic eyes complications | 3 years after intervention
  Using retinal photos and using the International Clinical Diabetic Retinopathy Disease Severity Scale
blood preassure | 3 years after intervention
  Blood pressure will be recorded with calibrated and validated electronic blood pressure equipment and appropriate sized cuff. Patients will sit in a chair in a quiet room for 5 minutes.
Lipids | 3 years after intervention
  Total cholesterol, low density lipoprotein, high density lipoprotein cholesterol and triglycerides will be measured

OTHER OUTCOMES:
health economics | from intervention and three years forward
  Direct healthcare resource consumption. Costs to Governments or Insurance companies plus private expenditure on health. Costs will include primary and secondary surgery, medication, laboratory tests, health provider reimbursement, private prescription charges and co-payments for medications
Quality of life score | three years after intervention
  Quality of life will be measured by the general health 36-item Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Thorell Anders, Professor, Principal Investigator — Karolinska Institutet
Locations (2):
- Ersta hospital, Stockholm, Stockholm County, Sweden
- St:Claraspital, Basel, Switzerland